CLINICAL TRIAL: NCT01656746
Title: Single Incision Laparoscopic Surgery (SILS) for Colorectal Disease - A Novel Approach
Brief Title: Single Incision Laparoscopic Surgery in Treating Patients With Colorectal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09123; NCI-2012-00604 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Adenomatous Polyp; Crohn Disease; Familial Adenomatous Polyposis; Hereditary Intestinal Polyposis Syndrome; Recurrent Colon Cancer; Stage I Colon Cancer; Stage IIA Colon Cancer; Stage IIB Colon Cancer; Stage IIC Colon Cancer; Stage IIIA Colon Cancer; Stage IIIB Colon Cancer; Stage IIIC Colon Cancer
Keywords: Colorectal Disease; SILS; colorectal surgery
MeSH Terms: conditions — Adenomatous Polyps; Crohn Disease; Adenomatous Polyposis Coli; Peutz-Jeghers Syndrome; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (single incision laparoscopic surgery) (Experimental): Patients undergo single incision laparoscopic surgery with GelPort® attachment.
  Interventions: Procedure: therapeutic laparoscopic surgery

INTERVENTIONS:
Procedure: therapeutic laparoscopic surgery — Undergo single incision laparoscopic surgery

SUMMARY:
This study is being done to evaluate single incision laparoscopic surgery (SILS) for colorectal diseases, compared to multi-port laparoscopic surgery. This study is also intended to standardize the SILS technique for colorectal diseases

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To report the experience of SILS procedure in the treatment of colorectal disease.

II. To standardize the SILS technique.

OUTLINE:

Patients undergo single incision laparoscopic surgery with GelPort® attachment.

After completion of study treatment, patients are followed up at 2 weeks, 3 and 6 months, and at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to give consent and comply with the evaluation and the treatment schedule
* Patients with disease processes limited to the right colon; this will include Crohn's disease, polyp disease, and cancers of the right colon
* American Society of Anesthesiologists (ASA) =< 3

Exclusion Criteria:

* Inability to obtain informed consent
* Previous right colon surgery
* Previous extensive abdominal surgery that would limit the laparoscopic approach
* Stage IV disease at surgery
* Metastatic disease diagnosed by computed tomography (CT), magnetic resonance imaging (MRI), or nuclear imaging
* Patient enrolled in other interventional study
* ASA score greater than 3
* Any condition which precludes compliance with the study (Investigator discretion)
* Co-morbid condition(s) that could limit the subject's ability to participate in the study or to comply with follow-up requirements, or that could impact the scientific integrity of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Operative time | Up to 1 year
  Summarized using descriptive statistics (i.e. means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data).
Length of skin and fascial incisions | Up to 1 year
  Summarized using descriptive statistics (i.e. means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data).
Estimated blood loss | Up to 1 year
  Summarized using descriptive statistics (i.e. means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data).
Oncologic sample including size of specimen removed, number of lymph nodes (LN) removed, pathological type and staging, lymph node, vessel or perineural invasion, and status of margins | Up to 1 year
  Summarized using descriptive statistics (i.e. means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data).

SECONDARY OUTCOMES:
Quality of life measured using the short form (SF)-12 health related quality of life scale (HQRL) scored using quality metric licensed software | Baseline
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Quality of life measured using the SF-12 HQRL scored using quality metric licensed software | 2 weeks
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Quality of life measured using the SF-12 HQRL scored using quality metric licensed software | 3 months
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Quality of life measured using the SF-12 HQRL scored using quality metric licensed software | 6 months
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue pain scale scored on the scale from 0 to 10 where 0 is no pain, and 10 is the maximum pain | Baseline
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue pain scale scored on the scale from 0 to 10 where 0 is no pain, and 10 is the maximum pain | 2 weeks
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue pain scale scored on the scale from 0 to 10 where 0 is no pain, and 10 is the maximum pain | 3 months
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue pain scale scored on the scale from 0 to 10 where 0 is no pain, and 10 is the maximum pain | 6 months
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue cosmesis scale scored on the scale from 0 to 10 where 0 is "worst scar", and 10 is the "best scar" | 2 weeks
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue cosmesis scale scored on the scale from 0 to 10 where 0 is "worst scar", and 10 is the "best scar" | 3 months
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.
Visual analogue cosmesis scale scored on the scale from 0 to 10 where 0 is "worst scar", and 10 is the "best scar" | 6 months
  Linear mixed model will be applied with repeated measures considering the observations from the same patient are correlated.

CONTACTS AND LOCATIONS:
Overall Officials: David Renton, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu